CLINICAL TRIAL: NCT01856296
Title: WINTHER: A Study to Select Rational Therapeutics Based on the Analysis of Matched Tumor and Normal Biopsies in Subjects With Advanced Malignancies
Brief Title: A Study to Select Rational Therapeutics Based on the Analysis of Matched Tumor and Normal Biopsies in Subjects With Advanced Malignancies
Acronym: WINTHER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2012-A01738-35; 2012/1946 (Other: CSET number)
Record Dates: First submitted 2013-05-15; First posted 2013-05-17 (Estimated); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Metastatic Cancer
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Experimental): ARM A patients with an identified oncogenic driver mutations/amplifications/translocations), who will potentially benefit from targeted therapies, either on the market or in clinical trials according to existing knowledge of matching oncogenic events with actionable drugs. This will be detected through Next Generation Sequencing (NGS) performed by Foundation Medicine, CLIA certified.
  Interventions: Procedure: Biopsy
- Arm B (Experimental): patients negative for oncogene events (which remains the majority), for whom genome based relevant information will be obtained through functional genomics (micro arrays and gene expression profiling) performed by Institut Gustave Roussy, and innovative computational methods enabling a rational choice of therapies. For such patients we will apply a new prediction model of efficacy of existing and under clinical trial drugs, based on differences in gene expression profiling between tumor and normal biopsies to be matched with relevant genes that are related to drug activities.
  Interventions: Procedure: Biopsy

INTERVENTIONS:
Procedure: Biopsy

SUMMARY:
An open non-randomized study using biology driven selection of therapies. WINTHER study will explore matched tumoral and normal tissue biopsies and will use a novel method for predicting efficacy of drugs. The aim is to provide a rational personalized therapeutic choice to all (100 %) patients enrolled in the study, harboring oncogenic events (mutations/ translocations/ amplifications, etc.) or not. The total number of patients treated in the study will be two hundred across all participating cancer centers (European countries -France; Spain-, Israel, USA and Canada). All centers will realize the same study independently.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Any histologic type of metastatic cancer, (except for lung and brain at US sites), in which histologic normal counterpart can be obtained.
* Progression by RECIST (Response Evaluation Criteria In Solid Tumors) or other criteria on at least one prior regimen for advanced disease.
* Ability to undergo a biopsy or surgical procedure to obtain fresh tumor biopsy paired with its normal counterpart.
* Age from 18 years
* Life expectancy of at least 3 months
* ECOG Performance status of 0 to 1
* Measurable or evaluable disease according to RECIST 1.1 criteria
* For U.S. sites, advanced cancer patients that have exhausted all effective therapy for their disease and have progressed after previous line of therapy (documented disease progression under last treatment received) and conventional methods of assigning new therapy would not be expected to increase survival by more than 3 months.

Exclusion Criteria:

* Any patient that might require a lung or brain biopsy are excluded (at US sites)
* Alteration of organ function or hematopoietic function as defined by the following criteria:

  1. Serum aspartate transaminase (AST) and serum alanine transaminase (ALT) >2.5 x upper limit of normal (ULN), except for patients with liver metastases, for which AST and ALT > 5.0 ULN is the exclusion criteria.
  2. Bilirubin > 2.0 ULN
  3. Polynuclear neutrophil < 1.5 x 109/L
  4. Platelets < 100 x 10 9/L
  5. Hemoglobin < 90 g/L
  6. Creatinine > 1.5 ULN
  7. Calcemia > 1.5 ULN
  8. Phosphatemia > 1.5 ULN
* Coagulation abnormality prohibiting a biopsy
* Symptomatic or progressive brain metastases detected by radio imaging, or meningeal
* Patient who received a personalized therapeutic treatment based on molecular anomaly during the treatment period prior to the WINTHER directed treatment (defining the PFS1). Hormonal therapy may be continued during WINTHER suggested therapy. The exclusion of prior matched targeted therapy includes but is not limited to all targeted therapeutics that are EMA approved and genomically matched to patients. If there are questions about whether or not a prior therapy is matched targeted treatment it will be agreed on by discussion between PIs who are also Clinical Management Committee members; the resolution should take place prior to starting WINTHER directed treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2013-04-23 (Actual); Primary Completion 2015-12-07 (Actual); Study Completion 2019-02-22 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | Up to 6 months
  To assess the individual outcome of patients with advanced malignancies, by comparing the progression-free survival (PFS) using a treatment regimen selected by a molecular analysis of a patient's tumor with the PFS for the most recent regimen on which the patient had experienced progression
  * ARM A : PFS2/PFS1 >1.5 in 50% of patients
  * ARM B : PFS2/PFS1 >1.5 in 40% of patients
  The primary endpoint of the study is the ratio of the PFS of the current treatment (PFS2) versus the previous treatment (PFS1). Because patients will be enrolled in the study while they are still on treatment (before progression), we expect that PFS for the previous treatment is fully observed. If patients withdrew from the treatment due to treatment related toxicity and lost to follow-up, it is considered that the PFS endpoint is reached. If patients are lost to follow up due to other reasons, PFS is censored at the time of last follow up.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Gustave Roussy, Villejuif, Val De Marne, France